CLINICAL TRIAL: NCT00342472
Title: Environmental and Biological Monitoring Pilot Study for Polycyclic Aromatic Hydrocarbons in Linxian, China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998008; OH98-C-N008
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Polycyclic Aromatic Hydrocarbons
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Two of the oldest individuals (a male and a female greater than 18 years of age) from each of 10-15 nonsmoking households from the high-risk region of Linxian, China

SUMMARY:
The overall goal of this project is to determine whether polycyclic aromatic hydrocarbons (PAHs) are contributing to the high rate of esophageal cancer in Linxian, China.

Esophageal cancer is one of the most fatal cancers worldwide with Linxian, China having one of the highest rates in the world. In the United States esophageal cancer causes approximately 10,000 deaths each year. It is the fourth most common cause of cancer death in black males and the eighth leading cause of cancer death in men of all races. Although several recent studies have identified some of the molecular changes associated with esophageal cancer, its prevention and treatment within high risk groups continues to be limited by our inability to identify specific etiologic agents.

Human exposure to PAHs, including benzo [a]pyrene (B[a]P), is associated with an increased rate of skin, lung, and upper GI tumors and also with an increased mortality from causes related to atherosclerosis. Evidence, including the preliminary results from histologic and food analysis pilot studies, supports the idea that this region's high rate of esophageal cancer may be related to long-term, high-level exposure to PAHs via inhalation of air-borne pollution and ingestion of food cooked with soft coal.

Thus, to assess the association of PAHs with the high rate of esophageal cancer in Linxian, China, we plan to analyze samples of food for the presence of PAHs, samples of blood for Hb adducts (a marker of long-term PAH exposure), samples of urine for 1-OH-Pyrene glucuronide (a maker of short-term PAH exposure), and samples of coal for characteristics that may be associated with increased carcinogenesis. We will also administer environmental questionnaires that will include questions about the type of fuel used for cooking and heating, the location and type of stove and/or heating unit (i.e., vented versus unvented), and time spent cooking.

DETAILED DESCRIPTION:
The overall goal of this project is to determine whether polycyclic aromatic hydrocarbons (P AHs) or acetaldehyde are contributing to the high rate of esophageal cancer in Linxian, China.

Esophageal cancer is one of the most fatal cancers worldwide and Linxian, China has some of the highest rates of this cancer in the world. In the United States esophageal cancer causes approximately 14,000 deaths each year. It is the fourth most common cause of cancer death in black males and the eighth leading cause of cancer death in men of all races. The prevention and treatment of esophageal cancer within high risk groups continues to be limited by our inability to identify specific etiologic agents.

Human exposure to PAHs, including benzo[a]pyrene (B [a]P) is associated with increased rates of skin, lung, esophageal and gastric tumors and also with an increased mortality from causes related to atherosclerosis. Preliminary results from histologic and food analysis pilot studies supports the possibility that the high rates of esophageal cancer in Linxian may be related to long-term, high level exposure to PAHs via inhalation of air-borne pollution and ingestion of food cooked with soft coal.

Exposure to acetaldehyde could also be an etiologically significant exposure in Linxian. Acetaldehyde is a carcinogenic metabolite, and small quantities of ethanol where recently found in homogenized Linxian food samples. The Salaspuro laboratory at the University of Helsinki has demonstrated that oral bacteria can produce acetaldehyde from food containing similar small concentrations of ethanol, so such acetaldehyde exposure could be etiologically significant in Linxian. Genetic polymorphisms, particularly those involving alcohol and acetaldehyde dehydrogenases, may also influence the effect of this exposure.

To assess the association of PAHs and acetaldehyde with the high rate of esophageal cancer in Linxian, China, we plant o analyze samples of food for the presence of PAHs, ethanol and acetaldehyde, samples of blood for Hb and DNA adducts( markers of long-term PAH or acetaldehyde exposure), samples of urine for 1-OH-Pyrene glucuronide (a marker of short term PAH exposure) samples of saliva for acetaldehyde and samples of coal for characteristics that may be associated with increased carcinogenesis. We will also administer environmental questionnaires that will include questions about the type of fuel used for cooking and heating, the location and types of stove and/or heating units, and the time spent cooking.

ELIGIBILITY:
* INCLUSION CRITERIA:

Two of the oldest individuals (a male and a female greater than 18 years of age) from each of 10-15 nonsmoking households from the high-risk region of Linxian, China and, to the extent that is possible, from appropriately age matched controls from a total of 20 nonsmoking individuals from the low-risk region of Gejiu, Yunnan province will be selected to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two of the oldest individuals (a male and a female greater than 18 years of age) from each of 10-15 nonsmoking households from the high-risk region of Linxian, China and, to the extent that is possible, from appropriately age matched controls from a total of 20 nonsmoking individuals from the low-risk region of Gejiu, Yunnan province will be selected to participate.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 1998-02-12 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
PAH exposure | single time point, when samples are collected
  To assess the association of PAHs and acetaldehyde with the high rate of esophageal cancer in Linxian, China, we plant to analyze samples of food for the presence of PAHs, ethanol and acetaldehyde,samples of blood for Hb and DNA adducts( markers of longterm PAH or acetaldehyde exposure), samples of urine for 1-OH-Pyrene glucuronide (a marker of short term PAH exposure) samples of salivafor acetaldehyde and samples of coal for characteristics that may be associated with increased carcinogenesis. We will also administer environmental questionnaires that will include questions about the type of fuel used for cooking and heating, the location and types of stove and /or heating units, and the time spent cooking.

CONTACTS AND LOCATIONS:
Overall Officials: Sanford M Dawsey, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Li JY. Epidemiology of esophageal cancer in China. Natl Cancer Inst Monogr. 1982;62:113-20. PMID 7167171
- [Background] Ronneberg A, Andersen A. Mortality and cancer morbidity in workers from an aluminium smelter with prebaked carbon anodes--Part II: Cancer morbidity. Occup Environ Med. 1995 Apr;52(4):250-4. doi: 10.1136/oem.52.4.250. PMID 7795740
- [Background] Mumford JL, He XZ, Chapman RS, Cao SR, Harris DB, Li XM, Xian YL, Jiang WZ, Xu CW, Chuang JC, et al. Lung cancer and indoor air pollution in Xuan Wei, China. Science. 1987 Jan 9;235(4785):217-20. doi: 10.1126/science.3798109.